CLINICAL TRIAL: NCT05363228
Title: The Effect of Tai Chi and Therapy by Dance and Movement on Blood Irisin Levels in Older Adults Over 65 Years of Age.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: University Hospital Vinohrady (Unknown); Faculty of Physical Education and Sport (Unknown)
Responsible Party: Principal Investigator, Hana Polanska, Researcher, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GAUK/268321
Record Dates: First submitted 2022-05-03; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Memory Deficits; Aging; Cognitive Impairment; Physical Activity; Mood Change
Keywords: Irisin; BDNF; Cognition; Aging; Therapy by Dance and Movement; Tai Chi
MeSH Terms: conditions — Memory Disorders; Cognitive Dysfunction; Motor Activity | interventions — Movement; Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Therapy by Dance and Movement (Experimental): Participants assigned to this part take part in Dance Movement Therapy twice a week (90 minutes each) for the duration of three months.
  Interventions: Behavioral: Therapy by Dance and Movement
- Control to Dance Movement Therapy (No Intervention): Participants assigned to this arm take part in no particular activity for the three months.
- Movement Therapy by Tai Chi (Experimental): Participants assigned to this part take part inTai Chi class twice a week (90 minutes each) for the duration of three months.
  Interventions: Behavioral: Tai Chi
- Control to Tai Chi (No Intervention): Participants assigned to this arm take part in no particular activity for the three months.

INTERVENTIONS:
Behavioral: Therapy by Dance and Movement — Therapy by dance and movement is based on the principals of movement-analysis by Rudolf Laban and Irmgard Bartenieff. Participants will attend sessions twice a week (90 minutes each) for the duration of three months.
  Arms: Therapy by Dance and Movement
Behavioral: Tai Chi — Tai Chi is based on somatic approach. Participants will attend sessions twice a week (90 minutes each) for the duration of three months.
  Arms: Movement Therapy by Tai Chi

SUMMARY:
The aim of this project is to estimate the effects of therapy with dance and movement and Tai Chi on irisin plasma levels, a myokine with proven neuroprotective effects, in the context of baseline levels of cognitive function and physical performance in seniors over 65 years of age.

It is empirically verified that physical activity can have a positive effect on cognitive function even in individuals with mild cognitive impairment. There may be a number of reasons why this is the case. Recently, research investigating the relationship between the secretion of certain myokines and their neuroprotective effects has gained importance. One of these myokines is irisin, which has recently been shown to have beneficial effects on the CNS by upregulating the expression of Brain Derived Neurotrophic Factor (BDNF) in the hippocampus in an animal model. Increased irisin levels as a consequence of exercise have recently been partially demonstrated in humans. What type of physical activity is most effective in terms of its effect on cognitive function in humans is another important scientific challenge. The possibility of influencing endocrine secretion of bioactive substances with proven effects on synaptic plasticity, neurogenesis and neuroprotection through effective therapies may help to combat neurodegenerative diseases, the prevalence of which is increasing with the average age of the population. According to Alzheimer's Disease International, 50 million people worldwide were affected by some form of neurodegenerative disease in 2017. The number of people affected is still rising. It is predicted that this number will reach 75 million sufferers by 2030 (https://www.alz.co.uk/research/statistics). Alzheimer's disease and multiple sclerosis are the two most common manifestations of neurodegenerative diseases. The effect of therapy with dance and movement and the effect of Tai Chi on blood irisin levels in the context of cognitive function and physical performance levels, has not yet been conclusively demonstrated.

DETAILED DESCRIPTION:
It is empirically verified that physical activity can have a positive effect on cognitive function even in individuals with mild cognitive impairment. There may be a number of reasons why this is the case. Recently, research investigating the relationship between the secretion of certain myokines and their neuroprotective effects has gained importance. One of these myokines is irisin, which has recently been shown to have beneficial effects on the CNS by upregulating the expression of Brain Derived Neurotrophic Factor (BDNF) in the hippocampus in an animal model. Increased irisin levels as a consequence of exercise have recently been partially demonstrated in humans. What type of physical activity is most effective in terms of its effect on cognitive function in humans is another important scientific challenge. The possibility of influencing endocrine secretion of bioactive substances with proven effects on synaptic plasticity, neurogenesis and neuroprotection through effective therapies may help to combat neurodegenerative diseases, the prevalence of which is increasing with the average age of the population. According to Alzheimer's Disease International, 50 million people worldwide were affected by some form of neurodegenerative disease in 2017. The number of people affected is still rising. It is predicted that this number will reach 75 million sufferers by 2030 (https://www.alz.co.uk/research/statistics). Alzheimer's disease and multiple sclerosis are the two most common manifestations of neurodegenerative diseases. The effect of therapy with dance and movement and the effect of Tai Chi on blood irisin levels in the context of cognitive function and physical performance levels, has not yet been conclusively demonstrated. The aim of this project is to estimate the effects of therapy with dance and movement and Tai Chi on irisin plasma levels, a myokine with proven neuroprotective effects, in the context of baseline levels of cognitive function and physical performance in seniors over 65 years of age.

Implementation of the project: the following personal data will be collected at the Consultation Room for Memory Disorders, AD Centrum Fakultní at the Královské Vinohrady Hospital (PPP AD FNKV): age, weight, height, sex, education, a brief medical history will be taken, current illness and current treatment will be determined, and a basic pharmacological and toxicological history will be taken. The probands who will be admitted to the experimental part of the project, based on the initial screening at the PPP AD FNKV, will have their cognitive function tested and 9 ml of venous blood drawn before and after the intervention at the PPP AD FNKV, and strength and physical performance tested at the UK FTVS. Thereafter, probands will be randomized to either the intervention groups or the control group. This randomized controlled trial will compare the effects of a movement and dance therapy based on Bartenieff fundamentals and the other type of intervention will be implemented as Tai Chi exercises. Both types of exercises are designed to place a greater emphasis on body perception, so that there is a connection between musculoskeletal coordination and movement in conjunction with an emotional experience focused on the ability to perceive bodily signals. This approach will activate cognitive functions more. The experimental part will be carried out with a time intensity of twice a week (90 min) for 12 weeks - all in two phases 09-2021 to 12-2021 and 09-2022 to 12-2022. The control group will be implemented on the principle of wait-list control group.

Characteristics of research participants: Based on the power analysis, we expect to recruit approximately 90 participants (age ≥ 65 - ≤ 80 years) from outpatients of the PPP AD FNKV and U3V UK FTVS participants, or other interested persons from Prague 6.

Individuals with advanced cognitive impairment, regular use of medications affecting cognitive performance, antidepressants, anxiolytics, and individuals with uncorrected hypertension and ischemic heart disease, acutee (especially infectious) disease, musculoskeletal disorders and chronic diseases limiting physical activity, as well as individuals in recovery after illness or injury cannot take part in the study.

Ethical aspects of research: The research will be conducted on seniors who will be enrolled in the research on the basis of voluntary informed consent. Since movement therapy has no negative side effects, it is an ethically conflict-free research from this perspective. On the other hand, a great benefit to society can be expected, in particular the development of a suitable exercise regimen that will be applicable to other age groups. Since the elderly are a specific and relatively easy to influence group, they will be adequately informed about the purpose of the research, and the benefits of the research for them and for the elderly population as a whole will be explained. Before signing the informed consent, the clarity and understanding of the information provided will be carefully checked.

ELIGIBILITY:
Inclusion Criteria:

* Is 65 years - 80 years in age
* His/her native language is Czech
* Is willing to visit the testing centre two times within 3-4 months
* Is willing to provide blood samples twice
* Is willing to take part in the movement therapy intervention
* is self-sufficient (handling finances, travelling without a chaperone, administration of medication, correct phone usage, filling forms, meal preparation)
* Has good vision; Can read and write, glasses are acceptable
* Has good hearing to hear and understand all instructions during examination
* Can walk well (walking aids are acceptable) to attend all the examinations and move well enough to take part in the movement therapy

Exclusion Criteria:

* Had been treated/Is currently being treated for the following psychiatric disorders: alcohol/medication/drug of abuse dependance, schizophrenia, psychotic disorder, bipolar disorder
* Had larger physical imparment which would interfere with the ability to take part in the Dance Movement and Tai Chi interventions
* Had severe neurological difficulties (epilepsy, stroke, severe head trauma, meningitis in the past 10 years, brain surgery, brain tumour, prolonged period(s) in an unconscious state - excluding general anaesthesia)
* Underwent a surgery/procedure under general anaesthesia in the past three years or has a planned procedure/surgery under general anaesthesia in the next 6 months over the course of this trial
* Is taking medication for depression or low mood

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in Irisin blood levels after 3 months of the intervention | baseline to 3 months
  Irisin levels measured from 9ml blood samples
Difference in Irisin blood levels between the arms at 3 months | 3 months
  Irisin levels measured from 9ml blood samples

SECONDARY OUTCOMES:
Change in brain derived neurotrophic factor (BDNF) levels at 3 months | baseline to 3 months
  BDNF measured from a 9ml blood samples.
Difference in brain derived neurotrophic factor (BDNF) levels at 3 months between the arms | 3 months
  BDNF measured from a 9ml blood samples.
Change from baseline cognitive function in the Amnesia Light and Brief Assessment (ALBA) at 3 months better outcome | baseline to 3 months
  ALBA is a validated measure assessing memory. The scale spans 0-12 points with higher number of points signifying better outcome
Difference in cognitive function in the Amnesia Light and Brief Assessment (ALBA) between the arms at 3 months | 3 months
  ALBA is a validated measure assessing memory. The scale spans 0-12 points with higher number of points signifying better outcome
Change from baseline cognitive function in Semantic word recollection (category: animals, 1 min) at 3 months | baseline to 3 months
  Semantic word recollection is a measure of cognitive function, results range from 0-cca 40, more points signify better outcome
Difference in cognitive function in Semantic word recollection (category: animals, 1 min) between the arms at 3 months | 3 months
  Semantic word recollection is a measure of cognitive function, results range from 0-cca 40, more points signify better outcome
Change in cognitive function in Semantic word recollection (category: letters, 1 min) at 3 months | baseline to 3 months
  Semantic word recollection is a measure of cognitive function, results range from 0-cca 40, more points signify better outcome
Difference in cognitive function in Semantic word recollection (category: letters, 1 min) at 3 months between the arms | 3 months
  Semantic word recollection is a measure of cognitive function, results range from 0-cca 40, more points signify better outcome
Change from baseline cognitive function in Rey Auditory Verbal Learning Test (RAVLT) at 3 months | baseline to 3 months
  RAVLT is a validated measure of cognitive function, it has 8 subscales, each of them ranging from 0-15, measured in raw scores which are connected to age-dependent population norm
Difference in cognitive function in Rey Auditory Verbal Learning Test (RAVLT) at 3 months between the arms | 3 months
  RAVLT is a validated measure of cognitive function, it has 8 subscales, each of them ranging from 0-15, measured in raw scores which are connected to age-dependent population norm
Change in baseline cognitive function in Wechsler Adult Intelligence Scale, Third edition (WAIS III) - "Symbols" subtest at 3 months | baseline to 3 months
  The WAIS III, subtest "Symbols" is a validated measure of cognitive function, the point scale ranges from 0-133 with larger point attainment signalling better outcome
Difference in cognitive function in Wechsler Adult Intelligence Scale, Third edition (WAIS III) - "Symbols" subtest at 3 months between the arms | 3 months
  The WAIS III, subtest "Symbols" is a validated measure of cognitive function, the point scale ranges from 0-133 with larger point attainment signalling better outcome
Change in baseline cognitive function in Trail Making Test (TMT), Parts A & B at 3 months | baseline to 3 months
  The TMT is a validated measure of cognitive function, the time upon completion is measured
Difference in cognitive function in Trail Making Test (TMT), Parts A & B at 3 months between the arms | 3 months
  The TMT is a validated measure of cognitive function, the time upon completion is measured
Change in the Clock Drawing Test at 3 months | baseline to 3 months
  A validated measure where participant is asked to draw a clock face with the time 23:20
Difference in the Clock Drawing Test at 3 months between the arms | 3 months
  A validated measure where participant is asked to draw a clock face with the time 23:20
Change in Line Picture Production test at 3 months | baseline to 3 months
  Participant is asked to produce as many as possible pictures consisting from 4 straight lines in 1 minute.
Difference in Line Picture Production test at 3 months between the arms | 3 months
  Participant is asked to produce as many as possible pictures consisting from 4 straight lines in 1 minute.
Change in Picture Naming and Immediate Recall test (PICNIR) at 3 months | Baseline to 3 months
  Cognitive measure where participants first write down names of 20 pictures and then are asked to recall these names within 1 minute
Difference in Picture Naming and Immediate Recall test (PICNIR) at 3 months between the arms | 3 months
  Cognitive measure where participants first write down names of 20 pictures and then are asked to recall these names within 1 minute.
Change in baseline mood in Geriatric Depression Scale at 3 months. | baseline to 3 months
  A self-report measure of mood, measured on 0-15 point scale, higher point attainment signifies worse outcome.
Difference in mood in Geriatric Depression Scale at 3 months. | 3 months
  A self-report measure of mood, measured on 0-15 point scale, higher point attainment signifies worse outcome.
Change from baseline self-sufficiency self-reported in Questionnaire of functional state (abbreviation in original language: subjective FAQ-CZ) at 3 months | baseline to 3 months
  FAQ-CZ is a self-report measure of self-sufficiency, it is measured on a scale of 0-30 with higher point attainment signalling worse outcome
Difference in self-sufficiency self-reported in Questionnaire of functional state (abbreviation in original language: subjective FAQ-CZ) at 3 months between the arms | 3 months
  FAQ-CZ is a self-report measure of self-sufficiency, it is measured on a scale of 0-30 with higher point attainment signalling worse outcome
Change in Sarcopenia at 3 months | baseline to 3 months
  An ultrasound imaging method for diagnosing sarcopenia based on changes in muscle geometric proportions: muscle thickness (MT), pennation angle (PA), fiber length (FL), and ultrasound sarcopenic index (USI) calculated as FL/MT.
Difference in Sarcopenia at 3 months between the arms | 3 months
  An ultrasound imaging method for diagnosing sarcopenia based on changes in muscle geometric proportions: muscle thickness (MT), pennation angle (PA), fiber length (FL), and ultrasound sarcopenic index (USI) calculated as FL/MT.
Change in knee extensor isometric strength and static fatigue at 3 months | baseline to 3 months
  Knee extensor isometric strength and static fatigue were measured by a stationary dynamometer: isometric torque (Nm), and fatigue index calculated as the Area Under Force vs. Time Curve of right knee extensor during a sustained 30 s maximal voluntary muscle contraction. Handgrip strength.
Difference in knee extensor isometric strength and static fatigue at 3 months between the arms | 3 months
  Knee extensor isometric strength and static fatigue were measured by a stationary dynamometer: isometric torque (Nm), and fatigue index calculated as the Area Under Force vs. Time Curve of right knee extensor during a sustained 30 s maximal voluntary muscle contraction. Handgrip strength.
Change in short physical performance battery (SPPB) at 3 months | baseline to 3 months
  The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests. It is used as a predictive tool for possible disability and can aid in the monitoring of function in older people.
Difference in short physical performance battery (SPPB) at 3 months between the arms | 3 months
  The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests. It is used as a predictive tool for possible disability and can aid in the monitoring of function in older people.
Change in Body Composition at 3 months | baseline to 3 months
  Body composition by a bioelectrical impedance analysis (BIA).
Difference in Body Composition at 3 months between the arms | 3 months
  Body composition by a bioelectrical impedance analysis (BIA).

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - Faculty Hospital Vinohrady, Prague
  - Faculty of Physical Education and Sport, Prague

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hola V, Polanska H, Jandova T, Jaklova Dytrtova J, Weinerova J, Steffl M, Kramperova V, Dadova K, Durkalec-Michalski K, Bartos A. The Effect of Two Somatic-Based Practices Dance and Martial Arts on Irisin, BDNF Levels and Cognitive and Physical Fitness in Older Adults: A Randomized Control Trial. Clin Interv Aging. 2024 Nov 6;19:1829-1842. doi: 10.2147/CIA.S482479. eCollection 2024. PMID 39525874